CLINICAL TRIAL: NCT06820125
Title: Isolated Versus Combined Cognitive and Motor High-tech Rehabilitation in Patients with Multiple Sclerosis
Brief Title: Isolated Versus Combined Cognitive and Motor High-tech Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Nicola Smania, MD, Clinical Professor, Doctor, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4257CESC
Record Dates: First submitted 2025-01-24; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-12

CONDITIONS: Rehabilitation; Multiple Sclerosis; Cognitive Deficit; Motor Deficits
Keywords: rehabilitation; multiple sclerosis; cognitive deficits; motor deficits
MeSH Terms: conditions — Multiple Sclerosis; Cognition Disorders; Neurologic Manifestations

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cognitive Group (CG) (Experimental): 60 minutes of cognitive training with a computerized device
  Interventions: Device: Cognitive rehabilitation: CG group
- Motor Group (MG) (Experimental): 60 minutes of robot-assisted gait training with the G-EO System
  Interventions: Device: Motor rehabilitation: MG group
- Combined Group (CbG) (Experimental): 30 minutes of cognitive training with a computerized device + 30 minutes of robot-assisted gait training with the G-EO System.
  Interventions: Device: Combined rehabilitation: CbG group

INTERVENTIONS:
Device: Cognitive rehabilitation: CG group — 60 minutes of cognitive training with a computerized device
  Arms: Cognitive Group (CG)
Device: Motor rehabilitation: MG group — 60 minutes of robot-assisted gait training with the G-EO System
  Arms: Motor Group (MG)
Device: Combined rehabilitation: CbG group — 30 minutes of cognitive training with a computerized device + 30 minutes of robot-assisted gait training with the G-EO System. To mitigate the effects of fatigue in sequential training, the patients included in this group will undergo the cognitive (treatment CG) and motor (treatment MG) sessions in a counterbalanced order (half of the participants will follow the CG-MG sequence, and the other half will follow the MG-CG sequence). Five-minute breaks will be provided between the cognitive and motor sessions.
  Arms: Combined Group (CbG)

SUMMARY:
The first aim of this project is to investigate the effects of different high-tech neurorehabilitation interventions (cognitive, motor, and combined cognitive-motor) on both cognitive and motor disability outcomes in people with multiple sclerosis (MS).

The second aim is to identify the cognitive and motor profiles of MS patients who benefit the most from either the combined cognitive-motor rehabilitation intervention or the isolated cognitive or motor treatments.

ELIGIBILITY:
Inclusion Criteria:

* presence of mild (one or two neuropsychological tests below the cut-off score, 5th percentile) or severe (more than two neuropsychological tests below the cut-off score, 5th percentile) cognitive impairment,
* mild to moderate walking disability with Expanded Disability Status Scale (EDSS) between 3 and 6,
* no relapse or associated steroid use in the past three months,
* adequate visual and auditory capacity to operate computer software.

Exclusion Criteria:

* presence of other neurological disorders than MS,
* major psychiatric disorders,
* high levels of anxiety and/or depression (score>20 for Depression scale and up to 14 for Anxiety scale on Italian adaptation of the Depression, Anxiety and Stress Scale (DASS-21),
* substance abuse,
* any type of rehabilitation intervention in the month prior to recruitment
* pharmacological therapy not well defined and/or changed during the study
* presence of paroxysmal vertigo
* lower limb botulinum toxin injections within the previous 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2026-07-05 (Estimated)

PRIMARY OUTCOMES:
Symbol Digit Modalities Test | The test is administered before the treatment, then after eight weeks of treatment, and finally two months after the end of the treatment
  This test evaluates the visual information processing speed and attention; the number of correct answers in 90 seconds is registered (higher scores indicate better performance).
2-minute walking test | The test is administered before the treatment, then after eight weeks of treatment, and finally two months after the end of the treatment
  The 2MWT will be administered to measure self-paced walking ability. Patients will be asked to walk back and forth, as fast as they could, along a 30-m indoor corridor in 2 minutes. No talking will be permitted during the test. The distance walked (in meters) will be recorded (higher scores indicated better performance).

SECONDARY OUTCOMES:
Brief Repeatable Battery (BRB) | The test is administered before the treatment, then after eight weeks of treatment, and finally two months after the end of the treatmen
  The the Brief Repeatable Battery (BRB) is composed of the Selective Reminding Test - SRT (to evaluate verbal learning and delayed memory recall; the words recalled in three different subtests are recorded); the Spatial Recall Test - SPART (to evaluate visuospatial learning and delayed memory recall; the total number of correct responses for the three trials and the delayed recall trial are recorded); the SDMT (described above); the Paced Auditory Serial Addition Test - PASAT (to assesses auditory information processing speed, attention, and calculation; the score is the sum of correct answers recorded - max 60); the Word List Generation -WLG (to assesses semantic verbal fluency; the score is the number of correct words recorded).
The Stroop Test (ST) | The test is administered before the treatment, then after eight weeks of treatment, and finally two months after the end of the treatmen
  The Stroop Test (ST), which evaluates attention and the ability to inhibit automatic responses. The Stroop effect is evaluated by computing a time interference effect (based on execution time) and an error interference effect (based on number of errors).
Trail Making Test (TMT) | The test is administered before the treatment, then after eight weeks of treatment, and finally two months after the end of the treatmen
  The Trail Making Test (TMT), which consists of two parts: the TMT-A, used as a measure of psychomotor speed and visual search/attention skills, and the TMT-B, used as a measure of attentional set-shifting and mental flexibility. Time needed to complete the tasks is recorded.
The Verbal Fluency Test (VF) | The test is administered before the treatment, then after eight weeks of treatment, and finally two months after the end of the treatmen
  The Verbal Fluency Test (VF), which is composed of 3 subtests: the Phonemic Fluency, the Semantic Fluency, and the Phonemic/Semantic Alternate Fluency test. For each trial, the number of correct words generated in 60 sec is recorded. Performance score in each subtest is the sum of the correct words generated in all trials.
The Modified Five Point Test (MFPT) | The test is administered before the treatment, then after eight weeks of treatment, and finally two months after the end of the treatmen
  The Modified Five Point Test (MFPT), which is a measure of figural fluency assessing the ability to initiate mental productivity and self-monitoring during a visual-spatial task. Performance is assessed by scoring the total number of correct and unique designs generated in 3 min (UDs), and the total number of UDs produced into strategies (CSs).
Test of Attentional Performance (TAP; version 2.3.1) | The test is administered before the treatment, then after eight weeks of treatment, and finally two months after the end of the treatmen
  The Test of Attentional Performance (TAP; version 2.3.1), which evaluates different aspects of attention; in particular, we will administer a Go/No-Go task, which examines the ability to perform an appropriate response under time pressure and to simultaneously inhibit an automatic behavioral response triggered by an external stimulus.
N-Back task | The test is administered before the treatment, then after eight weeks of treatment, and finally two months after the end of the treatmen
  The N-Back task be made up of a sequence of stimuli, and the task consists of indicating when the current stimulus matches the one from n steps earlier in the sequence. The load factor n can be adjusted to increase the task difficulty. We will administer the visual N-Back available from a computerized device.
Time up and Go (TUG) | The test is administered before the treatment, then after eight weeks of treatment, and finally two months after the end of the treatmen
  Time up and Go (TUG) will be administered to assess functional mobility of patients. In this test, patients have to stand up, walk 3 meters, turn around, walk back, and sit down. The time taken to complete the test is correlated with the level of functional mobility. Patients can perform the TUG also under a dual task condition in which they are required to count backwards from a randomly selected number between 20 and 100 while walking (TUG-COG). TUG-COG is considered a cognitive task because it investigates dual task ability.
  The TUG is a good general indicator of locomotor function, but the timed global performance does not provide any information regarding the mechanisms underlying the patient's disabilities and specific problems relating to each sub-task are not highlighted.
eight-infrared camera system (sampling frequency: 60-120 fps) with the VICON Vero 2.2 motion analysis system (Vicon Motion Analysis System Ltd), | The test is administered before the treatment, then after eight weeks of treatment, and finally two months after the end of the treatmen
  to specifically assess characteristics of gait, we will carry out gait analysis, which will be performed using an eight-infrared camera (sampling frequency of 60-120 fps) VICON Vero 2.2 motion analysis system (Vicon Motion Analysis System Ltd) synchronized with a two AMTI force plate. According to the Davis protocol, 16 reflective markers (14 mm diameter) will be positioned on the seventh cervical vertebra, the left and right anterior superior iliac spines (ASIS), the sacrum, the left and right mid-thighs, the left and right lateral femur condyles, the left and right mid-shanks, the left and right lateral malleoli, the dorsal aspect of the left and right feet (between the second and the third metatarsal head) and on the left and right calcanea [46]. Two analogue cameras will be integrated into the system and aligned with the sagittal and coronal planes. Gait cycle events (toe off and initial foot contact) will be defined automatically, using Vicon Clinical Manager software.
Modified Fatigue Impact Scale (MFIS) | The test is administered before the treatment, then after eight weeks of treatment, and finally two months after the end of the treatmen
  To evaluate the patients' fatigue we will provide the Modified Fatigue Impact Scale (MFIS), a 21-items shortened version of the 40-items Fatigue Impact Scale. Although no basic analyses of the MFIS have been published, it has been used in clinical practice and several clinical trials and intervention studies
The Multiple Sclerosis Quality of Life-29 (MSQOL-29) | The test is administered before the treatment, then after eight weeks of treatment, and finally two months after the end of the treatmen
  The Multiple Sclerosis Quality of Life-29 (MSQOL-29), the 29-items shortened version of the MSQOL-54, is a 29-item validated structured self-report questionnaire evaluating generic and MS-specific domains of health-related quality of life (QoL) in 7 multi-item subscales and 4 single-item subscales. Subscale scores are obtained by averaging the items within subscale and transforming the mean scores linearly to 0 to 100 possible scores. The higher the scores, the better the QoL. Physical Health Composite (PHC) and Mental Health Composite (MHC) are derived by combining scores of the subscales.
Client Satisfaction Questionnaire (CSQ-8) | At the end of the treatment
  a self-administered post-treatment questionnaire, comprised of eight items that evaluate the level of satisfaction regarding the care and quality of the service received and the level of fulfillment of the patient's expectations regarding the treatment administered. The total score of the questionnaire is 32 points, with higher values meaning higher satisfaction with the treatment received.

CONTACTS AND LOCATIONS:
Locations (1):
- Sezione medicina fisica e riabilitativa dipartimento di neuroscienze, Verona, verona, Italy